CLINICAL TRIAL: NCT00466479
Title: Topical Brimonidine vs Argon Laser Trabeculoplasty in Progressing Human Glaucoma. A Prospective Randomized Clinical Trial.
Brief Title: Brimonidine vs ALTP in Progressing Human Glaucoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Parma (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PARMANP001
Record Dates: First submitted 2007-04-26; First posted 2007-04-27 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Glaucoma
Keywords: neuroprotection; alpha one agonists; glaucoma; visual field
MeSH Terms: conditions — Glaucoma | interventions — Brimonidine Tartrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: brimonidine
Procedure: laser trabeculoplasty

SUMMARY:
This study is evaluating possible non-intraocular pressure (IOP) related effects of the alpha-1 agonist brimonidine in human subjects affected by a progressive glaucomatous optic neuropathy. Brimonidine was proven as neuroprotective in several pre-clinical animal studies.

DETAILED DESCRIPTION:
Patients with open angle glaucoma and a history of relative stability of the visual field are followed for 18 months. A visual field is measured every 3 months for a total number of n = 6 eligible fields at the end of this phase. Then, those eyes showing progression of the field (i.e. deterioration of th eexisting glaucoma), are randomized to receive either 0.2% brimonidine tartrate eyedrops b.i.d. or 360° argon laser trabeculoplasty in one session. Either treatment will be put "on top" of the pre-existing anti-glaucoma therapy. Then, a further 18-month phase is planned, with a sequnece of field taken at the same pace as the previous phase. Progression is detected (and measured) acording to a trend-analysis (i.e. regression vs time of single points and of clusters of adjacent points).

ELIGIBILITY:
Inclusion Criteria:

* Glaucomatous visual field defect on achromatic perimetry (24/2 Humphrey full threshold,abnormal GHT and CPSD, p<0.01) considered clinically "unstable"
* IOP < 20 mmHg on repeated readings with no more than 2 medications,
* Open angle on gonioscopy,
* Glaucomatous optic neuropathy (HRTII, Moorfields regression analysis),
* Clear lens (LOCS2 score < C1, N0, P0)
* Best corrected visual acuity better than 0.2 LogMAR (ETDRS chart),
* No previous bulbar surgery
* Manifest refraction within - 5 and + 2 diopters
* No comorbidity (AMD and diabetic retinopathy.and negative history for neurological diseases)

Exclusion Criteria:

* Closed angle
* Previous bulbar surgery
* Unstable IOP
* Unreliable visual fields on historic data

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 1999-08; Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
progression of visual field measured as loss of sensitivity in decibels per year
progression of visual field measured as number of eyes showing at least one cluster of points progressing

SECONDARY OUTCOMES:
number of drop out(s) for adverse events

CONTACTS AND LOCATIONS:
Overall Officials: stefano gandolfi, MD, Principal Investigator — University of Parma
Locations (1):
- sezione di Oftalmologia, Parma, Italy